CLINICAL TRIAL: NCT03844100
Title: Multi-center Single Sided Preliminary Study to Evaluate Effectiveness and Safety in Administrating CNU® Capsule to Refractory Functional Dyspepsia Patients
Brief Title: Effectiveness and Safety in Administrating CNU® Capsule to Refractory Functional Dyspepsia Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung III Jang, Assistant professor, MD, PhD, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2018-0300
Record Dates: First submitted 2018-12-11; First posted 2019-02-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Dyspepsia; Biliary Dysplasia
Keywords: Refractory Functional Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — 1-(2-chloroethyl)-1-nitrosourea; Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: single arm: patients with refractory functional dyspepsia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Refractory Functional Dyspepsia (Experimental): Patients with FD diagnosed by the Rome IV criteria, patients with Refractory Functional Dyspepsia
  * Person who have had early satiation and bothersome postprandial fullness for minimum 3 days a week and epigastric pain and epigastric soreness for minimum 1 day a week
  * Person with above symptoms that started at least 6 months before and continused for minimum 3 months
  * Person having no possible causes of above symptoms including organic disease, structural modification, systemic disease, and endocrinology-metabolic disease
  * Person who do not respond to at least 2 general treatments for FD
  * Dyspepsia symptoms that can disrupt daily life (global overall symptom scale score =>5)
  Interventions: Drug: efficacy and safety of CNU® Capsule

INTERVENTIONS:
Drug: efficacy and safety of CNU® Capsule — All subjects take 250mg CNU capsule orally 1 capsule per time, 2 times a day (morning, evening / at meal or after meal) for 12 weeks.
  Other Names: CNU® Capsule (Trihydrated magnesium salt of kenodeoxycholic acid and ursodeoxycholic acid, 250 mg)

SUMMARY:
Refractory Functional Dyspepsia (FD) means a state that no symptom was improved in spite of appropriate treatment for the FD.

It may be challenging to discriminate the symptoms of FD from the symptoms of bile dyspepsia resulting from the biliary system. As the bile dyspepsia may induce epigastralgia as with functional dyspepsia and both imaging medical tests and blood tests show normal findings, it is difficult to discriminate it from the FD with only these tests.

Thus this study intends to perform a therapeutic use clinical study for efficacy and safety on symptom improvement by administrating CNU capsule to the patients with RFD.

DETAILED DESCRIPTION:
Functional Dyspepsia means a pain or discomfort of epigastrium originated from the stomach or duodenum without any causative organic or metabolic disease. For its standard criteria, "Rome IV diagnosis criteria" was used, where more than on symptoms including bothersome postprandial fullness, early satiation, epigastric pain, and epigastric soreness should have been elicited at least 6 months before and continued for at least 3 months in total.

Refractory Functional Dyspepsia means a state that no symptom was improved in spite of appropriate treatment for the functional dyspepsia.

The pathogenesis of Functional Dyspepsia has not been fully identified yet. Its standard therapies include prokinetics, analgesics, H2-receptor antagonists, proton pump inhibitors, antacids, serotonin receptor antagonists, proton pump inhibitors, antacids, serotonin receptor antagonists, and antidepressants. As these therapies has lower efficacy and drug related adverse reactions, the RFD patients who do not respond to medication need another therapeutic option.

It may be challenging to discriminate the symptoms of FD from the symptoms of bile dyspepsia resulting from the biliary system. As the bile dyspepsia may induce epigastralgia as with functional dyspepsia and both imaging medical tests and blood tests show normal findings, it is difficult to discriminate it from the FD with only these tests.

Therefore even though the epigastralgia or upper abdominal discomfort met the Rome IV criteria for the FD, the possibility that it, in part was actually resulted from the bile dyspepsia cannot be eliminated.

The CNU capsule is a choleretic used for bile dyspepsia as a complex agent of trihydrated magnesium salt of kenodeoxycholic acid and ursodeoxycholic acid, which are being marketed.

Thus this study intends to perform a therapeutic use clinical study for efficacy and safety on symptom improvement by administrating CNU capsule to the patients with RFD.

ELIGIBILITY:
Inclusion Criteria:

1. Person over 19 years old as of the date of submission
2. Among patients with FD diagnosed by the Rome IV criteria, patients with RFD

   * Person who have had early satiation and bothersome postprandial fullness for minimum 3 days a week and epigastric pain and epigastric soreness for minimum 1 day a week
   * Person with above symptoms that started at least 6 months before and continused for minimum 3 months
   * Person having no possible causes of above symptoms including organic disease, structural modification, systemic disease, and endocrinology-metabolic disease
   * Person who do not respond to at least 2 general treatments for FD
   * Dyspepsia symptoms that can disrupt daily life (global overall symptom scale score =>5)
3. Persons who submitted written consent to participate in this study

Exclusion Criteria:

1. Patient with biliary disease other than bile stone, scraps in the gall and bile tract, and polyps of gallbladder
2. Patient with structurally abnormal biliary system from congenital malformation or other reasons
3. Patients with endocrinology-metabolic disease that can affect mobility of gastrointestinal tract and biliary system such as diabetes and abnormal thyroid function
4. Patient who cannot discontinue any drug that can provoke abdominal symptoms
5. Patient with disease or damage in central nervous system (cerebral hemorrhage and cerebral infarction with residual disorder) and autonomic nervous system (vertebrate)
6. Patient with renal disorder and electrolyte imbalance
7. Patient who received gastrointestinal surgery (excluding appendectomy and hemorrhoidectomy)
8. Patient with frequent biliary colic or infection of biliary infection
9. Obstructive jaundice patient
10. Severe renal disease patient
11. Patient with variceal bleeding, hepatic coma, ascites, and needs for acute liver transplantation
12. Patient with severe pancreatic disease
13. Person scheduled to receive combined administration of below drugs:

    * Drug with considerable hepatic toxicity Antacid agent containing cholestyramine, medical charcoal, magnesium and aluminum hydroxide
    * alpha-methydopa
    * Drug to increase bile secretion of cholesterol ( estrogen, hormonal contraception agent, partial lipid lowering agent), drug to reduce blood cholesterol
14. Patient with hypersensitivity to this drug or any component of this drug
15. Patient with severe biliary obstruction
16. Patient with radiopaque, calcificated bile stone
17. Patient with acute cholecystitis
18. Patient with peptic ulcer
19. Patient with coloenteritis like Crohn disease
20. Cholestasis patient
21. Patient with abnormality in gallbladder contraction (below 40% of GB ejection fraction)
22. Person relevant to below criteria, as results of tests conducted in screening

    * Person with BUN exceeding 3 times of normal upper limit
    * Person with blood creatinine exceeding 3 times of normal upper limit
    * Person with total bilirubin exceeding 3 times of normal upper limit
    * Person with direct bilirubin exceeding 3 times of normal upper limit
    * Person with AST(sGOT) and ALT(sGPT) exceeding 3 times of normal upper limit
    * Person with ALP(alkaline phosphatase) exceeding 3 times of normal upper limit
    * Person with GGT(gamma-glutamyl transferase) exceeding 3 times of normal upper limit
23. Woman who is pregnant or lactating and women in childbearing age who uses no reliable contraceptive measure or doesn't agree to keep contraception during pregnancy period
24. Person who cannot understand purpose and methods of this study such as mental patients or patients with drug and alcohol abuse
25. Other persons considered by any investigator to have some difficulties in performing this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Improvement of symptoms | 12weeks after CNU capsules
  The primary outcome variable will be the percentage of subjects to report that they are improved or unchanged or deteriorated or No assessable in overall symptoms compared to baseline on a 7-point Global Overall Symptom Scale (GOS). The GOS is assessed on a 7-point scale, with the severity scale from 1 (Normal, not at all ill) through to 7 (Among the most severely ill patients).

SECONDARY OUTCOMES:
The Total Number of subjects Experiencing at Least one Adverse Event During the study | for 12 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - CHA Bundang Medical Center, Seongnam, Bundang-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - In Ha University Hospital, Incheon, Jung-gu
  - Soon Chun Hyang University Hospital, Cheonan, Cheonan, Namdong-gu
  - Gachon University Gil Medical Center, Incheon, Namdong-gu

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available untill all patients are enrolled and be open to all researchers for 1 year
Access Criteria: Only researchers.